Official Title of the study: Effects of Intermittent Fasting in Metabolic Dysfunction **Associated Fatty Liver Disease** 

NCT number: NCT06664684

Date of the document: 06.05.2022

Written Inform Consent

In this study, we will evaluate the effects of dietary modification and dietary time modification on biochemical parameters, fatty liver and liver damage levels in adults with

metabolic dysfunction-associated fatty liver disease.

If you agree to participate in this study, a questionnaire form including your sociodemographic characteristics, information about your lifestyle, 3-day food consumption record and food consumption frequency will be applied to you. Participants will be asked to follow a specially prepared diet programme for 8 weeks. In addition, anthropometric measurements (height, body weight, body fat-muscle analysis, waist circumference, hip circumference) will be taken and necessary biochemical analyses will be performed with blood samples taken from you. Thus, it is aimed to reveal the effect of diet therapy on the disease. The study has no risk and side effects for the participants. The results obtained from the study will contribute to improvements and developments

We encourage you to participate in this study. Participation in the study is voluntary. This means that you are free to take part in this study or not. You will not be asked for any remuneration for taking part in this study, nor will you receive any remuneration for taking part in the study. The results of the research can be published in scientific environments and used in student education, provided that your name remains confidential. Make your decision after reading and understanding the information about the study. If your decision is positive after reading this information, please sign the form.

in the nutritional programmes of Metabolic Dysfunction Associated Fatty Liver Patients.

I have read the text above, which shows the information that should be given to the volunteer before the study. I have been given written and verbal explanations about these. Under these conditions, I agree to participate in this clinical trial voluntarily and without any pressure or coercion.

Name-surname and signature of the volunteer:

Name, surname and signature of the researcher who made the explanations: